CLINICAL TRIAL: NCT03480724
Title: Assessing the Efficacy of Virtual Reality Analgesia (VRA) in Pediatric Patients for Pain Control During Botox Injections for Spasticity Management: A Randomized Control Trial
Brief Title: Assessing the Efficacy of Virtual Reality Analgesia (VRA) in Pediatric Patients for Pain Control
Acronym: PEDSPAINVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite efforts no additional participants were able to be enrolled since March 2020.
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Academy of Physical Medicine and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-6501
Record Dates: First submitted 2017-04-14; First posted 2018-03-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 3 groups of patients One group with no VR One group with Oculus rift VR One group with google cardboard box VR
Who Masked: Outcomes Assessor
Masking Description: The outcome accessor will have no patient contact and will not have access to the information on the type of intervention study patients were given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Google Cardboard VRA (Active Comparator): This group of subjects will receive VRA intervention using Google Cardboard Virtual reality head- mounted display powered by a iPod touch.
  Interventions: Other: Google Cardboard VRA
- Oculus Rift VRA (Active Comparator): This group of subjects will receive VRA with Oculus Rift
  Interventions: Other: Oculus Rift VRA
- Control (No Intervention): This group of subjects will receive no intervention beyond standard sedation, anesthetic, and/or restraint-this group will serve as the control group

INTERVENTIONS:
Other: Google Cardboard VRA — Intervention was randomized and shuffled.
  Arms: Google Cardboard VRA
Other: Oculus Rift VRA — Intervention was randomized and shuffled.
  Arms: Oculus Rift VRA

SUMMARY:
To evaluate the efficacy of virtual reality analgesia (VRA) for pediatric patients undergoing Botulinum toxin injections (BTI) for spasticity management. Patients will be assigned to one of three groups; one group of subjects will randomly be assigned to VRA intervention using Google Cardboard Virtual reality head- mounted display powered by a iPod touch, a second group of subjects will receive VRA with Oculus Rift, and a third group of subjects will receive no intervention beyond standard sedation, anesthetic, and/or restraint-this group will serve as the control group.

DETAILED DESCRIPTION:
Group 1: Oculus Rift This group will receive BTI's per conventional protocols. They will wear the Oculus Rift VRHMD (Figure

1) powered by the laptop pc (Figure 2) during the procedure viewing a VR 360 degree video of their choice. Measurements in pain and anxiety will be taken per the outcome measures listed above.

Group 2: Google Cardboard VRHMD This group will receive BTI's per conventional protocols. They will wear the Google cardboard VRHMD (Figure 3) powered by iPod touch/smartphone (Figure 4) during the procedure viewing a VR 360 degree video of their choice. Measurements in pain and anxiety will be taken per the outcome measures listed above.

Group 3. Control This group will receive BTI's per conventional protocols without VRA intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children with spasticity requiring BTI
* Children ages 5 - 18
* Children who have contraindications for sedation for BTI
* Children with intact vision who can attend VR intervention

Exclusion Criteria:

* Children who have uncontrolled seizures > than 4 per year
* Children who are not attentive to VR secondary to poor concentration, poor cognition to external stimuli
* Children on different treatments for spasticity such as baclofen pump, phenol block. For patients who receive phenol block, phenol block will be held during the visits with VR intervention to avoid confounding results
* Children with poor bleeding control
* Children who request general anesthesia/IV sedation.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Severity of Pain Measurement | About 20 minutes per patient.
  Measurement of pain using the Face Legs Activity Cry Consolability scale (FLACC scale) which is a Behavioral Pain Assessment Scale. Each category is scored on the 0-2 scale, that results in total score of 0-10.
  0= Relaxed and comfortable , 1-3 = Mild discomfort, 4-6=Moderate pain, 7-10= Severe discomfort or pain or both. Lower score is a good outcome and higher score is a bad outcome. The assessment is for all the subjects in the study.

SECONDARY OUTCOMES:
Measurement of severity of anxiety | About 20 minutes per patient
  Measurement of anxiety using Short State-Trait Anxiety Inventory (STAI) Anxiety scale which is a self-evaluation questionnaire completed by the patient's parent or guardian about how they feel and how the child feels at that moment.
  It consists of 6 questions each having scale 1-4. 1 being Not at all and 4 being Very much. The questions are as follows:
  1. I feel calm
  2. I am tense
  3. I feel upset
  4. I am relaxed
  5. I feel content
  6. I am worried

CONTACTS AND LOCATIONS:
Overall Officials: Yuxi Chen, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- E-MMC - Rehabilitation Medicine, The Arthur S. Abramson Department of, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No